CLINICAL TRIAL: NCT05178459
Title: Withings Study to Analyse the Accuracy of Screening Small Fiver Neuropathy With a Bathroom Scale
Acronym: WISUDO
Status: Completed | Type: Observational
Sponsor: Withings (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021-A02624-37
Record Dates: First submitted 2021-12-15; First posted 2022-01-05 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Neuropathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetic: Patient diagnosed with diabetes
  Interventions: Diagnostic Test: Neuropathy measurement
- Neuropathic without diabetes: Patient diagnosed with neuropathy without diabetes
  Interventions: Diagnostic Test: Neuropathy measurement

INTERVENTIONS:
Diagnostic Test: Neuropathy measurement — Patient will step on Withings WBS08 and on the Sudoscan to get their sudomotor dysfunction caused by the neuropathy evaluated.

SUMMARY:
The aim of this study is to evaluate the diagnostic performance of Withings WBS08 to screen small fiber neuropathy.

DETAILED DESCRIPTION:
Patients with neuropathy are included in hospitals. Each patient will have his neuropathy evaluated with Withings WBS08 and its reference the Sudoscan.

ELIGIBILITY:
Inclusion Criteria:

* The subject is an adult, man or woman (18 years old or more)
* Subjects affiliated or eligible to a social security system
* Subjects having expressed their consent to take part in the study
* Two type of patients are included in the study :

  * Patients having diabetes (80% of the inclusion)
  * Non diabetic patients having a lower limbs neuropathy (20% of the inclusion)

Exclusion Criteria:

* Minors under 18 years old
* Subject is pregnant or trying to get pregnant
* Subjects having a pacemaker
* Subjects having refused to give their consent
* Vulnerable subjects according to the French regulation in force:

  * Individuals deprived of liberty by a court, medical or administrative order
  * Individuals legally protected or unable to express their consent to take part in the study
  * Individuals unaffiliated to or not beneficiary of a social security system
  * Individuals who fit in multiple categories above
* Individuals linguistically or mentally unable to express their consent
* Individuals having an lower limb amputation bigger than toes
* Individuals not able to stand still for a few minutes
* Individuals under antidepressant medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In and out patients from endocrinology and neuropathy departments
Sampling Method: Non-Probability Sample
Enrollment: 177 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2022-08-08 (Actual)

PRIMARY OUTCOMES:
Sudomotor dysfunction diagnostic performance evaluation | 10 months
  The diagnostic performance of the Withings WBS08 will be established using the sensitivity and the specificity for an electrochemical skin conductance threshold (moderate dysfunction and severe dysfunction).

SECONDARY OUTCOMES:
Evaluate the accuracy of Withings WBS08 to measure the sudomotor function on each foot and by averaging the value on both feet. | 10 months
  The root-mean-square error (RMSE) and the mean absolute error (MAE) between the sudomotor function value measured by the Withings WBS08 and the Sudoscan as reference on each foot and by averagin g both feet.
Compare the diagnostic of Withings WBS08 to diabetes neuropathy questionnaires | 10 months
  The correlation between diabetes neuropathy questionnair es and Withings WBS08.
Safety use of this device | 10 months
  The rate of adverse effects.

CONTACTS AND LOCATIONS:
Overall Officials: Louis Potier, Dr, Principal Investigator — Bichat-Claude Bernard Hospital
Locations (4):
- France (4):
  - Henri-Mondor Hospital, Créteil, Île-de-France Region
  - Lariboisière Hospital, Paris, Île-de-France Region
  - Cochin Hospital, Paris, Île-de-France Region
  - Bichat-Claude Bernard Hospital, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Riveline JP, Mallone R, Tiercelin C, Yaker F, Alexandre-Heymann L, Khelifaoui L, Travert F, Fertichon C, Julla JB, Vidal-Trecan T, Potier L, Gautier JF, Larger E, Lefaucheur JP. Validation of the Body Scan(R), a new device to detect small fiber neuropathy by assessment of the sudomotor function: agreement with the Sudoscan(R). Front Neurol. 2023 Oct 31;14:1256984. doi: 10.3389/fneur.2023.1256984. eCollection 2023. PMID 38020587